CLINICAL TRIAL: NCT03828474
Title: Sickness Evaluation at Altitude With Acetazolamide at Relative Doses
Acronym: SEAWARDII
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carrie Jurkiewicz, Clinical Instructor, Department of Emergency Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 49724
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-02

CONDITIONS: Acute Mountain Sickness
Keywords: acetazolamide; chemoprophylaxis; altitude
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Visually identical pills
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Acetazolamide 125mg twice daily (Experimental): Acetazolamide pill 125mg twice daily by mouth, started the night prior to ascent and continued for 3 total doses
  Interventions: Drug: Acetazolamide Pill
- Acetazolamide 62.5mg twice daily (Experimental): Acetazolamide pill 62.5mg twice daily by mouth, started the night prior to ascent and continued for 3 total doses
  Interventions: Drug: Acetazolamide Pill

INTERVENTIONS:
Drug: Acetazolamide Pill — Acetazolamide pill
  Other Names: Diamox

SUMMARY:
The specific aim of this study is to evaluate whether acetazolamide 125mg daily is no worse than acetazolamide 250mg daily in decreasing the incidence of acute mountain sickness (AMS) in travelers to high altitude. The study population is hikers who are ascending at their own rate under their own power in a true hiking environment at the White Mountain Research Station, Owen Valley Lab (OVL) and Bancroft Station (BAR), Bancroft Peak, White Mountain, California

DETAILED DESCRIPTION:
Acute mountain sickness (AMS) is a constellation of symptoms including headache, sleep disturbance, fatigue, dizziness, and nausea, vomiting, or anorexia that commonly occurs in travelers ascending to altitudes above 2,500m. AMS incidence varies based on altitude and ascent profile with rates reported from 25 to 75% in tourists, trekkers, and mountaineers at North American altitudes. Symptom onset is typically six to twelve hours after arrival at high altitude. This self-limited disease can be debilitating when severe, and left unrecognized or untreated may progress to potentially fatal high altitude cerebral edema (HACE). While gradual ascent has proven effective in preventing AMS, this approach is often impractical to recreationists, search and rescue, disaster relief, and military operations.

Acetazolamide increases minute ventilation by 10-20% in subjects at altitude, and hastens acclimatization. It is well established that acetazolamide's main site of action is in the kidney, where it generates a metabolic acidosis through renal bicarbonate wasting and attenuates the effects of hypoxemic-induced respiratory alkalosis. Recommended dosing of acetazolamide for AMS prophylaxis has significantly decreased since early days of use in the 1960s. The current recommended dose of acetazolamide for this indication is 125 mg twice daily, as opposed to historical recommendations of 500mg or 750mg daily. Multiple meta-analyses have concluded that when compared with higher doses, 250mg of acetazolamide daily has been shown to be equally efficacious, with the added benefit of decreasing side effects including paresthesias and dysgeusia. A randomized controlled trial confirmed effectiveness of acetazolamide 125mg twice daily in prevention of AMS when started prior to ascent. In this study, it was found that 125mg twice daily corresponded to a range of 3-5mg/kg/day, depending on subject weight. Within this range, those on the lower dosing range did not have a greater incidence or severity of AMS. For subjects weighing between 50kg (110 lbs) - 83kg (183 lbs), a dose of 250mg/day acetazolamide would fall in this range. Interestingly, mountaineers and trekkers have anecdotally reported protection against AMS with 125mg/day of acetazolamide, a dose below 3-5mg/kg for anyone over 41kg (91lb).

Finding the lowest effective dose of acetazolamide for AMS prophylaxis is important because side effects of this medication can mimic AMS, decreasing the specificity of disease scoring on the validated Lake Louise Questionnaire (LLQ) and subsequent AMS diagnosis and chemoprophylactic effectiveness.Keeping in mind that LLQ is scored based on symptoms of headache, gastrointestinal symptoms, fatigue and weakness, and dizziness and lightheadedness, whatever effect acetazolamide has on AMS prevention may be obscured by its side effects that mimic the very same disease. Falsely positive LLQ scores in trekkers and mountaineers taking acetazolamide prophylaxis may lead to unnecessary pharmacologic treatment or even evacuation. From the perspective of high altitude research, participants randomized to or already taking acetazolamide may skew study results by decreasing LLQ specificity and potentially leading researchers to overestimate incidence of AMS.

ELIGIBILITY:
Inclusion Criteria:

* Able to complete moderate hike at altitude
* Live at elevation < 4,000 ft
* Able to arrange own transportation to study site
* Available for full study duration (Friday night - Sunday morning)

Exclusion Criteria:

* Pregnancy
* Slept at altitude > 4,000 ft within 1 week of study
* Allergy to acetazolamide or sulfa drugs
* NSAIDs, acetazolamide, or corticosteroids within 48 hours prior to study start
* History of severe anemia, severe heart disease, advanced COPD/emphysema or sickle cell disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Incidence of acute mountain sickness | 2 days
  Incidence of acute mountain sickness by Lake Louise Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Jurkiewicz, MD, Principal Investigator — Stanford University
Locations (1):
- White Mountain Research Center, Bishop, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Patot MC, Leadbetter G 3rd, Keyes LE, Maakestad KM, Olson S, Hackett PH. Prophylactic low-dose acetazolamide reduces the incidence and severity of acute mountain sickness. High Alt Med Biol. 2008 Winter;9(4):289-93. doi: 10.1089/ham.2008.1029. PMID 19115912
- [Background] Leaf DE, Goldfarb DS. Mechanisms of action of acetazolamide in the prophylaxis and treatment of acute mountain sickness. J Appl Physiol (1985). 2007 Apr;102(4):1313-22. doi: 10.1152/japplphysiol.01572.2005. Epub 2006 Oct 5. PMID 17023566
- [Background] Hackett PH, Roach RC. High-altitude illness. N Engl J Med. 2001 Jul 12;345(2):107-14. doi: 10.1056/NEJM200107123450206. No abstract available. PMID 11450659
- [Derived] Lipman GS, Jurkiewicz C, Burnier A, Marvel J, Phillips C, Lowry C, Hawkins J, Navlyt A, Swenson ER. A Randomized Controlled Trial of the Lowest Effective Dose of Acetazolamide for Acute Mountain Sickness Prevention. Am J Med. 2020 Dec;133(12):e706-e715. doi: 10.1016/j.amjmed.2020.05.003. Epub 2020 May 29. PMID 32479750